CLINICAL TRIAL: NCT05929417
Title: Feasibility of a Benzodiazepine Deprescribing Intervention in Older Adults Living in the Belgian Community Setting
Brief Title: Benzodiazepines Deprescribing in the Community Setting: Intervention Feasibility
Acronym: END-IT CS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Collaborators: EBPracticenet (Unknown); Fonds National de la Recherche scientifique (FNRS) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CLIP/2023/01
Record Dates: First submitted 2023-05-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Benzodiazepine Deprescribing
Keywords: Benzodiazepines; Deprescribing; Community setting; Older adults

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- END-IT intervention for the community setting (Experimental): The community pharmacist will distribute an educational brochure to the patient. He will also propose to the patient to communicate about a potential benzodiazepine deprescribing with his/her general practitioner through a document called pharmaceutical proposal.
  Interventions: Other: END-IT intervention for the community setting
- Control (No Intervention): The participants will receive the usual care. The community pharmacists allocated to the control group will have access to the intervention material at the end of the study.

INTERVENTIONS:
Other: END-IT intervention for the community setting — The intervention was described in the arm/group descriptions.
  Arms: END-IT intervention for the community setting

SUMMARY:
The goal of this feasibility study is to evaluate the feasibility of an intervention, led by the pharmacist, aiming at benzodiazepines and z-drugs deprescribing in older adults living in the Belgian community setting. The main questions it aims to answer are:

* To what extent will Belgian community pharmacists adhere to the intervention?
* To what extent will patients and general practitioners take up the intervention to deprescribe benzodiazepines and z-drugs?
* To what extent is the design of the recruitment and data collection process feasible and acceptable for all participants?

Participants will receive an educational brochure from their pharmacist. Their pharmacist will also propose to send a new standardized form to their general practitioner to enhance collaboration about a potential benzodiazepine deprescribing.

Researchers will compare this intervention to usual care to see if the intervention is feasible and to gather first data on intervention effectiveness in benzodiazepine deprescribing.

ELIGIBILITY:
Inclusion Criteria:

* being aged ≥65 years,
* taking a benzodiazepine receptor agonist for ≥4 weeks (Anatomical Therapeutic Chemical codes: N05BA, N05CD, N05CF and N03AE01)
* being a regular patient of the community pharmacy (defined as ≥ 4 visits/12 previous months).

Exclusion Criteria:

* Severe mental illness (assessed through having an active prescription of any antipsychotic medication).
* Dementia or significant cognitive impairment (assessed through an active prescription or any past prescription during the last 12 months of anticholinesterase inhibitors or memantine) and/or pharmacist's judgment).
* Patients unable to read or communicate in French.
* Ongoing benzodiazepine receptor agonist withdrawal at the time of recruitment.
* Known current alcohol withdrawal.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Pharmacists' adherence to the intervention | At 3 months
  Has the intervention been implemented as intended? (e.g: global number of implemented intervention components)
Pharmacists' adherence to the intervention | At 6 months
  Has the intervention been implemented as intended? (e.g: global number of implemented intervention components)
Participants' responsiveness | At 3 months
  How far participants (pharmacists, patients, and general practitioners) have responded to the intervention and have been engaged by the intervention: e.g. number of altered prescriptions).
Participants' responsiveness | At 6 months
  How far participants (pharmacists, patients, and general practitioners) have responded to the intervention and have been engaged by the intervention: e.g. number of altered prescriptions).
Feasibility of the recruitment process | At 6 months
  The feasibility of the recruitment will be assessed (e.g. the ratio between the number of included patients and patients contacted for participation).
Feasibility of the data collection process | At 6 months
  The feasibility of the data collection process will be assessed through the quality of the collected data (rate of missing data).

SECONDARY OUTCOMES:
Contextual factors potentially influencing the intervention effects at the patient-level. | At baseline
  Use of a questionnaire to assess factors that could explain potential differences in intervention implementation between patients.
Contextual factors potentially influencing the intervention effects at the pharmacist-level. | At baseline
  Use of a questionnaire to assess factors that could explain potential differences in intervention implementation between pharmacies.
Mechanisms of impact potentially influencing the intervention | At baseline
  Use a questionnaire to assess mechanisms of impact in relation with how the intervention is supposed to have its effects.
Mechanisms of impact potentially influencing the intervention | At 3 months
  Use of a questionnaire to assess mechanisms of impact in relation with how the intervention is supposed to have its effects.
Mechanisms of impact potentially influencing the intervention | At 6 months
  Use of a questionnaire to assess mechanisms of impact in relation with how the intervention is supposed to have its effects.
Exploratory benzodiazepine deprescribing rate analysis | At 3 months
  Defined as benzodiazepine reduction or cessation at 6 months
Exploratory benzodiazepine deprescribing rate analysis | At 6 months
  Defined as benzodiazepine reduction or cessation at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Spinewine, PhD, Principal Investigator — UCLouvain, Louvain Drug Research Institute/Clinical pharmacy research group
Locations (1):
- UCLouvain, Woluwe-Saint-Lambert, Belgium

IPD SHARING:
Plan to Share IPD: No
Only publishable project data relating to the main analysis and research output will be shared on a data repository after an embargo period of 2 years after June 2024. All relevant documentation necessary to facilitate data re-use will be shared along with the datasets.

REFERENCES:
- [Derived] Petein C, Chevallereau T, Aikpitanyi J, Evrard P, Tubeuf S, Henrard S, Spinewine A. Protocol to evaluate the feasibility of the D-PRESCRIBE intervention adapted to the Belgian community setting (END-IT CS study). BMJ Open. 2025 Mar 4;15(3):e085434. doi: 10.1136/bmjopen-2024-085434. PMID 40037665